CLINICAL TRIAL: NCT07149818
Title: A Single-arm Phase 2 Prospective Clinical Study of Linprixel in the Treatment of Relapsed/Refractory Autoimmune Hemolytic Anemia
Status: Not yet recruiting | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Chen Miao, Peking Union Medical College Hospital, Peking Union Medical College Hospital
Other Study IDs: Linperlisib-AIHA
Record Dates: First submitted 2025-06-11; First posted 2025-09-02 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Autoimmune Hemolytic Anemia
Keywords: Autoimmune Hemolytic Anemia
MeSH Terms: conditions — Anemia, Hemolytic, Autoimmune | interventions — parsaclisib

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- parsaclisib 40mg qd
  Interventions: Drug: Parsaclisib

INTERVENTIONS:
Drug: Parsaclisib — parsaclisib 40mg qd

SUMMARY:
wAIHA or EVANS syndrome: Linpriril 40mg, oral, once daily. The therapeutic effect will be evaluated after 4 weeks. If the therapeutic effect does not reach the PR, the dose will be increased to 60mg once a day. After continuing to take it for 4 weeks, the therapeutic effect will be evaluated again. If the PR is not reached, it can be increased to 80mg. If the PR is still not reached after continuing to take it for 4 weeks, it will be discontinued (for a total of 12 weeks). The initial dose is 40mg, taken orally once a day. If the therapeutic effect reaches PR or above after 4 weeks, continue taking this dose. The evaluation is the same as before every 4 weeks. The research period was 12 weeks. The duration of continuous treatment for effective patients is determined by the researchers, and the dosage of the drug can be reduced or increased.

cAIHA: Linpriril 80mg, oral administration, once daily. The therapeutic effect was evaluated every 4 weeks. The research period was 12 weeks. The treatment was discontinued if the therapeutic effect did not reach the PR within 12 weeks. The duration of continuous treatment for effective patients is determined by the researchers, and the dosage of the drug can be reduced or increased.

ELIGIBILITY:
Inclusion Criteria:

（1）Age ≥18 years old (2) Clearly diagnosed wAIHA or EVANS syndrome, cAIHA, primary or secondary connective tissue diseases. If it is secondary, there are no indications for the treatment of connective tissue diseases involving other systems.

(3) Patients who relapse or are refractory after at least two lines of treatment (previous treatments include glucocorticoids, CD20 monoclonal antibodies or at least two other immunosuppressants). Refractory is defined as the failure to achieve partial remission after 3 months of stable dose treatment with immunosuppressants.

(4) hb≤100 g / L (5) Those with complete clinical data, high treatment compliance, and those who have signed the informed consent form; (6) If glucocorticoids are being taken, they should be discontinued or the minimum maintenance dose has been taken for at least two weeks, and the minimum maintenance dose (≤15mg/day) should be continued subsequently (7) The infusion of CD20 monoclonal antibody should be at least 3 months or more. If the stable dose of immunosuppressants such as cyclosporine and sirolimus has been taken for at least 3 months, they should be discontinued upon enrollment.

Exclusion Criteria:

1. Those with incomplete functions of organs such as the heart, liver and lungs; Patients with acute renal insufficiency
2. Combined with connective tissue diseases, other vital organs are involved.
3. Uncontrolled infection or bleeding after standard treatment. Standard treatment for uncontrolled active infections of HIV, HCV or HBV.
4. Combined with advanced uncontrolled malignant tumors and lymphomas.
5. At the time of screening, the subjects had other types of uncorrected anemia, such as nutritional anemia, etc
6. Pregnant or lactating women.
7. Those who have used PI3Kδ inhibitors within the past 6 months;
8. Those who have participated in other clinical trials within three months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Record complete demographic data, improve the patient's medical history and physical examination.
  2. Routine examinations include blood routine (including reticulocytes), biochemistry (liver and kidney function, lactate dehydrogenase, ferritin, folic acid, vitamin B12), coagulation function, direct anti-human globulin test (DAT) and typing, colagglutinin test, autoantibody, antiphospholipid antibody, immunoglobulin, serum protein electrophoresis, and TB cell subset analysis. Cytokines (flow cytometry), chest and abdominal CT or abdominal ultrasound.
  3. Bone Marrow smear, biopsy, flow immunotyping, chromosome (optional)
Sampling Method: Non-Probability Sample
Enrollment: 22 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
The overall response rate (ORR) at 12 weeks | 12 weeks
  The overall response rate (ORR)
The complete response rate (CRR) at 12 weeks | 12 weeks
  The complete response rate (CRR) at 12 weeks

SECONDARY OUTCOMES:
The incidence of adverse events | 12 weeks
  The incidence of adverse events

IPD SHARING:
Plan to Share IPD: No